## Woebot for Substance Use Disorders

## NCT04096001

## Statistical Analysis Plan

Descriptive statistics (means and frequencies) will be used to describe the sample and examine program feasibility and acceptability ratings. Change scores (pre- minus post-treatment) will be calculated and bivariate correlations will be used to examine associations between changes in substance use (i.e., AUDIT-C scores, DAST-10 scores, and substance use occasions), as well as confidence, depression, and anxiety scores. T-tests will be conducted to examine changes from pre- to post-treatment in substance use, confidence, mood and pain by participants' current therapy and psychiatric medication status.